CLINICAL TRIAL: NCT05027373
Title: A Randomized, Double-blind, Placebo-controlled Parallel Trial of Safety, Tolerability and Pharmacokinetic of Recombinant Anti-IL-1β Humanized Monoclonal Antibody by Single Subcutaneous Injection in Healthy Subjects
Brief Title: Safety, Tolerability and Pharmacokinetic of Recombinant Anti-IL-1β Humanized Monoclonal Antibody Injection
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunshine Guojian Pharmaceutical (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SSGJ-613-HH-I-01
Record Dates: First submitted 2021-08-17; First posted 2021-08-30 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Systemic Juvenile Idiopathic Arthritis; Periodic Fever Syndrome
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SSGJ-613 (Experimental)
  Interventions: Drug: SSGJ-613
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SSGJ-613 — SSGJ-613 injection is 200mg/2mL solution in a single vial.The solution is a clear to slightly opalescent, colorless to a slightly yellow tint.
  Arms: SSGJ-613
Drug: Placebo — Placebo injection is 2mL excipient solution in a single vial.The solution is clear and colorless.
  Arms: Placebo

SUMMARY:
This study is Safety, Tolerability and Pharmacokinetic of Recombinant anti-IL-1β Humanized Monoclonal Antibody injection in Healthy Subjects. Pharmacokinetics, Pharmacodynamics and Anti-drug antibody (ADA) data will be collected; Drug safety, tolerability and immunogenicity for healthy subjects will be evaluated.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled parallel trial of safety, tolerability and pharmacokinetic of Recombinant anti-IL-1β Humanized Monoclonal Antibody by single subcutaneous injection with five different doses in healthy subjects. There are 5 groups as follows: 0.03mg/kg (S1), 1.0mg/kg (S2), 3.0mg/kg (S3), 6.0mg/kg (S4) and 10.0mg/kg (S5); and 2 subjects were included in the S1 group (both received study drugs); 8 subjects were included in each of the S2 ~ S5 groups (of which 6 received study drugs and 2 received placebo). In each group, two subjects were sentinels (1 received the study drug and 1 placebo). Pharmacokinetics, Pharmacodynamics and Anti-drug antibody (ADA) data will be collected; Drug safety, tolerability and immunogenicity for healthy subjects will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Chinese healthy participants, male or female, aged 18 to 45 (including both ends)
* The body mass index (BMI) is in the range of 19.0~28.0 kg•m-2 (including both ends), and the weight of men is generally not less than 50kg, while the women is generally not less than 45kg
* Male participants and their partners or female participants must agree to take one or more non-drug contraceptives (such as complete abstinence, contraceptive rings, partner ligation, etc.) , and there is no sperm donation or egg donation plan until 3 months after finished the study
* Participants should fully understand the purpose, nature, methods and possible adverse reactions of the trial, volunteer to participate in the trial and sign the informed consent
* Participants could communicate well with the researchers and compliance with the trial

Exclusion Criteria:

* Those who are allergic to the study drug and any of its excipients. Subjects who have a history of allergy to monoclonal antibodies
* Subjects who have or are currently suffering from any serious clinical diseases 3-6 months before screening, such as circulatory system, endocrine system, nervous system, digestive system, respiratory system, urogenital system, hematology, immunology, psychiatry and metabolic abnormalities or any other that can interfere with the study results
* Clinical laboratory examinations (blood routine, urine routine, blood biochemistry, coagulation function, etc.), auxiliary examinations (chest X-ray, abdominal ultrasound) found to be abnormal and have clinical significance
* Positive for Hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HbcAb), anti- Hepatitis C virus antibodies (HCV), or anti-human immunodeficiency virus (HIV)
* Alcoholics or frequent drinkers within 3 months before the trial, drinking more than 14 units per week (1 unit alcohol ≈360 mL beer or 45 mL spirits or 150 mL wine), or those who have a positive alcohol breath test (screening period or baseline period) or couldn't prohibit alcohol during the trial
* Those who smoked more than 5 cigarettes per day during the 3 months before screening, or have a positive urine nicotine screening test (screening period or baseline period)
* Drug abusers or those who have used soft drugs (such as marijuana) within 3 months or took hard drugs (such as cocaine, phencyclidine, etc.) within 1 year before the trial, or have positive drug abuse screening (morphine, Ketamine, tetrahydrocannabinol acid, methamphetamine , dimethyldioxyamphetamine, cocaine)
* Has taken any prescription medicine, non-prescription medicine, Chinese patent medicine within 14 days before administration
* Has received any monoclonal antibody drugs within 3 months before administration
* Has a history of vaccination within 3 months before dosing, or intend to receive vaccines during the study
* Was previously enrolled in other clinical trials within 3 months before dosing
* Blood donors or subjects who lost a lot of blood (> 400 mL, except for women's physiological period) or those who received blood transfusion or used blood products within 3 months
* Can't tolerate venipuncture or has a history of halo needles and halo blood
* Has known or suspected pregnancy or lactation
* Abnormal vital signs (SBP <90 mmHg or ≥140 mmHg, DBP <55 mmHg or ≥90 mmHg; heart rate <50 bpm or> 100 bpm; body temperature <35.4℃ or > 37.3℃) or abnormal ECG (QTcF ≥450 ms) or physical examination are clinically significant (according to the judgment of clinical research doctors)
* Those who are infected and need to be treated for acute or chronic infections, as follows:

  * Suffering from herpes zoster within 12 months before screening;
  * Currently in any inhibitory treatment for chronic infections (eg, tuberculosis, pneumocystis, cytomegalovirus, herpes simplex virus, herpes zoster virus, and atypical mycobacteria);
  * A history of tuberculosis or contact with patients with open tuberculosis in the past 6 months,or a T-spoT-positive results;
  * Infected with parasites within 3 months before administration;
  * Hospitalized for infectious diseases within 30 days before administration;
  * Received anti-infective drugs (including antibacterial, antiviral, antifungal, or antiparasitic drugs) by parenteral administration (iv or im) 30 days before administration
* Subjects who are unsuited to the study for any reason, judged by the investigators

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2021-08-13 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Cmax | up to 112 days
Tmax | up to 112 days
AUC0-t | up to 112 days
t1/2 | up to 112 days
CL/F | up to 112 days
Vd/F | up to 112 days
Ke | up to 112 days
AUC0-∞ | up to 112 days
AE | up to 112 days
SAE | up to 112 days

SECONDARY OUTCOMES:
total IL-1β | up to 112 days
free IL-1β | up to 112 days
ADA | up to 112 days
  Bridging method will be used to detect the incidence and titer for ADA through one three-step detection strategy, that is preliminary screening, confirmation and titer

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Xuhui District Central Hospital, Shanghai, Shanghai Municipality, China